CLINICAL TRIAL: NCT05691699
Title: A Phase 1 First in Human, Single and Multiple Ascending Dose and Food Effect and Drug-Drug Interaction in Healthy Subjects to Evaluate the Safety, Tolerability and Assessment of Pharmacokinetics of ABBV-903
Brief Title: A Study to Assess Adverse Events and How Single and Multiple Ascending Doses of ABBV-903 Move Through the Body in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M24-112
Record Dates: First submitted 2023-01-09; First posted 2023-01-20 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Healthy Volunteer
Keywords: ABBV-903
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Part 1, ABBV-903 (Experimental): Participants will receive a single ascending dose of ABBV-903 in Part 1.
  Interventions: Drug: ABBV-903
- Part 1, Placebo (Experimental): Participants will receive a single ascending dose of placebo in Part 1.
  Interventions: Drug: Placebo for ABBV-903
- Part 2, ABBV-903 (Experimental): Participants will receive multiple ascending doses of ABBV-903 in Part 2.
  Interventions: Drug: ABBV-903
- Part 2, Placebo (Experimental): Participants will receive multiple ascending doses of placebo in Part 2.
  Interventions: Drug: Placebo for ABBV-903
- Part 3, Sequence 1 (Experimental): Participants in Part 3 will follow Sequence 1.
  Interventions: Drug: ABBV-903; Drug: Itraconazole
- Part 3, Sequence 2 (Experimental): Participants in Part 3 will follow Sequence 2.
  Interventions: Drug: ABBV-903; Drug: Itraconazole

INTERVENTIONS:
Drug: ABBV-903 — Capsule; oral
  Arms: Part 1, ABBV-903; Part 2, ABBV-903; Part 3, Sequence 1; Part 3, Sequence 2
Drug: Placebo for ABBV-903 — Capsule; oral
  Arms: Part 1, Placebo; Part 2, Placebo
Drug: Itraconazole — Capsule; oral
  Arms: Part 3, Sequence 1; Part 3, Sequence 2

SUMMARY:
The purpose of this study is to evaluate adverse events and tolerability of single and multiple doses of ABBV-903, and to assess how the drug moves through the body in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) is => 18.0 to <= 32 kg/m2 after rounded to the nearest tenth, at Screening and upon initial confinement.
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile and a 12-lead electrocardiogram (ECG).

Exclusion Criteria:

* History of any clinically significant illness/infection/major febrile illness, hospitalization, or any surgical procedure within 30 days prior to the first dose of study drug.
* History of epilepsy, any clinically significant cardiac, respiratory (except mild asthma as a child), renal, hepatic, gastrointestinal, hematologic or psychiatric disease or disorder, or any uncontrolled medical illness.
* Evidence of dysplasia or history of malignancy (including lymphoma and leukemia) other than successfully treated non-metastatic cutaneous squamous cell, basal cell carcinoma or localized carcinoma in situ of the cervix.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2023-10-23 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Baseline to Day 36
  Cmax will be assessed.
Time to Cmax (Tmax) | Baseline to Day 36
  Tmax will be assessed.
Apparent Terminal Phase Elimination Constant (β) | Baseline to Day 36
  Apparent terminal phase elimination constant (β) will be assessed.
Terminal Phase Elimination Half-life (t1/2) | Baseline to Day 36
  Terminal phase elimination half-life (t1/2) will be assessed.
Area Under the Plasma Concentration-time Curve (AUC) | Baseline to Day 36
  AUC will be assessed.
Area Under the Plasma Concentration-time Curve from Time 0 Until the Last Measurable Concentration (AUCt) | Baseline to Day 36
  AUCt will be assessed.
Area Under the Plasma Concentration-time Curve from Time 0 Until Infinity (AUCinf) | Baseline to Day 36
  AUCinf will be assessed.
Number of Participants with Adverse Events (AEs) | Baseline to Day 66
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Acpru /Id# 251279, Grayslake, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.abbvieclinicaltrials.com/study/?id=M24-112